CLINICAL TRIAL: NCT06256965
Title: Left Ventricular Ejection Fraction and Oxidative Stress Markers in Patients Subjected to Car-diac Surgery With Cardiopulmonary Bypass
Brief Title: Cardiopulmonary Bypass and Ventricular Remodeling
Acronym: CBP-VR
Status: Completed | Type: Observational
Sponsor: University of Chile (Other)
Collaborators: Hospital del Salvador (Other)
Responsible Party: Principal Investigator, RODRIGO CASTILLO, Rodrigouch, University of Chile
Other Study IDs: CBA180619
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Atrial Fibrillation; Heart Failure
Keywords: left ventricular ejection fraction; oxidative stress; cardiopulmonary bypass; atrial tissue
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure | interventions — Lipid Peroxidation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Biospecimen Retention: Samples Without DNA — 1. Tissue from right atrial appendage were obtained at surgical time after sternotomy and froozen at -80 Celsius degrees.
  Whoole blood samples obtained at surgical time after sternotomy were centrifuged at 3000 × g for 10 min. Plasma samples from each patient were stored at -80°C until performing the biochemical determinations of oxidative stress status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with present reduced left ventricular ejection fraction: patients with preoperatively shows in echocardiographic parameters LVEF lower 40%.
  Interventions: Diagnostic Test: Detection of peri-operative atrial fibrillation
- patients with present preserved left ventricular ejection fraction: patients with preoperatively shows in echocardiographic parameters LVEF higher 40%.
  Interventions: Diagnostic Test: Detection of peri-operative atrial fibrillation

INTERVENTIONS:
Diagnostic Test: Detection of peri-operative atrial fibrillation — atrial tissue and plasma from patients with atrial fibrillation detection were analyzed for determine lipid and protein oxidation, and detect markers of myocardial injury.
  Other Names: Detection of oxidative stress markers of protein and lipid peroxidation

SUMMARY:
The goal of this observational study is determine if reduced ventricular ejection fraction is a factor that determines a pro-oxidant imbalance in patients subjected to cardiac surgery with cardiopulmonary bypass.

The main questions are:

* 1. Preoperative reduced left ventricular function determines higher blood and atrial tissue oxidative stress in patients subjected to cardiopulmonary bypass
* 2. Oxidative stress markers in atrial tissue of cardiac surgical patients with develop atrial fibrillation The main tasks participants will be asked to do is register the symptoms of arrhythmia and heart failure. Also, obtain a electrocardiographic register if any present palpitations or chest pain with clinical significance This study not present a comparison group.

DETAILED DESCRIPTION:
1. Atrial fibrillation detection: continuous ECG monitoring was performed 24 to 48 h after CBP. Whenever arrhythmia symptoms occurred, a 12-lead ECG was performed every 12 h for 5 days. The presence of ECG-documented atrial fibrillation for at least 1 min was considered as a postoperative atrial fibrillation event.
2. Samples and Biopsies: All patients were subjected to the same surgical procedure, including the same induction and anesthesia protocol, and the execution by the same medical team. Surgical access was via a median sternotomy incision, and all anastomoses were sutured by hand. Protection of myocardial tissue was accomplished with crystalloid cold potassium cardioplegic solution. In cardiac surgery, at the time of pericardiocentesis, samples of right appendage (approximately 200mg) were obtained immediately before starting extracorporeal circulation. They were immediately frozen in liquid nitrogen and stored at -80°C. Blood samples were collected in chilled vacutainers containing 4 mM disodium EDTA and centrifuged at 3000 × g for 10 min. Plasma samples from each patient were stored at -80°C until performing the biochemical determinations.
3. Pre-operative Echocardiographic images: All echocardiographic analyses were performed at the Echocardiography Unit of the National Thorax Institute using GE Vivid E9 equipment at the baseline visit (7 days before surgery). The strain analyses were performed using a semi-automated speckle tracking technique (EchoPAC, GE Medical Systems, Milwaukee, Wisconsin) using a model of the entire LV (the 3 apical views). Inadequately tracked segments were excluded. A 3D full-volume acquisition of the LV using a matrix array transducer with the highest possible volume rate was be attempted in all patients. LV volumes and LVEF were measured offline (3DLVQ, EchoPAC, GE Medical Systems, Milwaukee, Wisconsin), with an abnormal LVEF identified as <40 %.
4. Biochemical parameters of oxidative stress. Determinations in plasma and atrial tissue samples (obtained during cardiac surgery, at the time of pericardiocentesis) and treated under the same experimental conditions.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years, chronic heart failure (WHO-functional class II, III) for at least 3 months before surgery. At the baseline visit, 7-10 days before surgery, the patients were classified by echocardiography as HF with pLVEF (LVEF >40%) or HF with rLVEF (LVEF ≤40%).

Exclusion Criteria:

* Patients with history or evidence of AF, previous myocardial infarction, current use of amiodarone, severe congestive heart failure (New York Heart Association class III or IV), presence of prosthetic valves, congenital valvular disease, chronic rheumatic, neoplastic diseases, liver insufficiency, severe chronic kidney disease (serum creatinine >2.5 mg/dl), recent infections ( 2 weeks) and emergency surgery or repair of cyanotic heart disease.

In addition, patients receiving nonsteroidal anti-inflammatory drugs, corticosteroids, antioxidants, vitamins, or fish oil supplements, three months before surgery were also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A prospective study was conducted in patients referred to the Cardiac Surgery De-partment from the National Thoracic Institute from Santiago, Chile, between October to December 2021, inclusively. The follow-up includes 2 groups: i) patients with preserved LVEF (pLVEF, n=7) and ii) patients with reduced LVEF (rLVEF, n=5).
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2022-06-13 (Actual)

PRIMARY OUTCOMES:
Postoperative atrial fibrillation | cardiac recording monitoring from surgery until the fifth postoperative day
  The presence of ECG-documented atrial fibrillation for at least 1 min was considered as a postoperative atrial fibrillation event.

SECONDARY OUTCOMES:
Oxidative stress markers | Samples obtained at surgical time and on fourty eight hours from surgery
  Tissue and plasma lipid peroxidation were measured as TBARS and 8-isoprostanes levels. Nitrotyrosine levels were detect in atrial tissue from show an oxidation of proteins

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, University of Chile, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Noubiap JJ, Sanders P, Nattel S, Lau DH. Biomarkers in Atrial Fibrillation: Pathogenesis and Clinical Implications. Card Electrophysiol Clin. 2021 Mar;13(1):221-233. doi: 10.1016/j.ccep.2020.10.006. PMID 33516400
- [Result] Thavendiranathan P, Negishi T, Somerset E, Negishi K, Penicka M, Lemieux J, Aakhus S, Miyazaki S, Shirazi M, Galderisi M, Marwick TH; SUCCOUR Investigators. Strain-Guided Management of Potentially Cardiotoxic Cancer Therapy. J Am Coll Cardiol. 2021 Feb 2;77(4):392-401. doi: 10.1016/j.jacc.2020.11.020. Epub 2020 Nov 18. PMID 33220426
- [Result] Benzie IF, Strain JJ. The ferric reducing ability of plasma (FRAP) as a measure of "antioxidant power": the FRAP assay. Anal Biochem. 1996 Jul 15;239(1):70-6. doi: 10.1006/abio.1996.0292. PMID 8660627
- [Result] Szymczyk G, Beltowski J, Marciniak A, Kotarski J. Serum isoprostanes levels in patients after abdominal hysterectomy. Rocz Akad Med Bialymst. 2005;50:322-4. PMID 16358993
- [Result] Gutierrez-Camacho LR, Kormanovski A, Del Carmen Castillo-Hernandez M, Guevara-Balcazar G, Lara-Padilla E. Alterations in glutathione, nitric oxide and 3-nitrotyrosine levels following exercise and/or hyperbaric oxygen treatment in mice with diet-induced diabetes. Biomed Rep. 2020 May;12(5):222-232. doi: 10.3892/br.2020.1291. Epub 2020 Mar 11. PMID 32257185
- [Result] Farias JG, Herrera EA, Carrasco-Pozo C, Sotomayor-Zarate R, Cruz G, Morales P, Castillo RL. Pharmacological models and approaches for pathophysiological conditions associated with hypoxia and oxidative stress. Pharmacol Ther. 2016 Feb;158:1-23. doi: 10.1016/j.pharmthera.2015.11.006. Epub 2015 Nov 23. PMID 26617218
- [Result] Xu Y, Guo W, Zeng D, Fang Y, Wang R, Guo D, Qi B, Xue Y, Xue F, Jin Z, Li Y, Zhang M. Inhibiting miR-205 Alleviates Cardiac Ischemia/Reperfusion Injury by Regulating Oxidative Stress, Mitochondrial Function, and Apoptosis. Oxid Med Cell Longev. 2021 Jun 29;2021:9986506. doi: 10.1155/2021/9986506. eCollection 2021. PMID 34306321
- [Result] Farias JG, Molina VM, Carrasco RA, Zepeda AB, Figueroa E, Letelier P, Castillo RL. Antioxidant Therapeutic Strategies for Cardiovascular Conditions Associated with Oxidative Stress. Nutrients. 2017 Sep 1;9(9):966. doi: 10.3390/nu9090966. PMID 28862654